CLINICAL TRIAL: NCT00530114
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel Group, Fixed Dose Study of AMG 223 in Subjects With Chronic Kidney Disease on Hemodialysis With Hyperphosphatemia
Brief Title: Study to Assess Fixed Dosing of AMG 223 in Subjects With Chronic Kidney Disease on Hemodialysis With Hyperphosphatemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20070664
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: End Stage Renal Disease; Chronic Kidney Disease; Hyperphosphatemic; Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): 1.0 g TID orally 3.0 g TID orally 4.0 g TID orally 5.0 g TID orally
  Interventions: Drug: Placebo
- AMG 223 (Experimental): 1.0 g TID orally 3.0 g TID orally 4.0 g TID orally 5.0 g TID orally
  Interventions: Drug: AMG 223

INTERVENTIONS:
Drug: AMG 223 — 1.0 g TID orally 3.0 g TID orally 4.0 g TID orally 5.0 g TID orally
  Arms: AMG 223
Drug: Placebo — 1.0 g TID orally 3.0 g TID orally 4.0 g TID orally 5.0 g TID orally
  Arms: Placebo

SUMMARY:
The primary objectives of this study are the following:

1. To demonstrate that AMG 223 will produce a statistically significant reduction in serum phosphorus compared with placebo over a 3 week treatment period in subjects with CKD receiving dialysis
2. To describe a dose response for AMG 223
3. To evaluate the safety and tolerability of AMG 223

ELIGIBILITY:
Inclusion Criteria:

* Maintenance hemodialysis 3 times a week for at least 3 months prior to screening
* Single pool Kt/V at least 1.2 or urea reduction ratio at least 65%
* Serum phosphorus level of 3.5 to 6.5 mg/dL inclusive at screening
* No change(s) in type or dose of non-investigational phosphate binder(s) for at least 1 month prior to screening
* Serum albumin > 3.0 mg/dL at screening
* If applicable, an increase in serum phosphorus of greater than or equal to 1.5 mg/dL, and a serum phophorous level > 5.5 mg/dL and less than or equal to 10 mg/dl during the washout period
* If applicable, stable doses (defined as no change in dose for at least 1 month prior to screening) of Vitamin D replacement, calcimimetic agents, or bedtime calcium supplements
* Willingness to avoid intentional changes in diet such as fasting or dieting

Exclusion Criteria:

* Previous intolerance leading to discontinuation of polymer-based phosphate binder therapy
* History of noncompliance with phosphate binder therapy in the opinion of the investigator
* Anticipating or scheduled for a living related-donor kidney transplant, or a prior recipient of a kidney transplant
* Current use of antiarrhythmic or anti-seizure medication
* Active ethanol or drug dependence or abuse, excluding tobacco use
* A screening serum calcium (corrected for albumin) < 8.4 mg/dL
* History of bowel obstruction, swallowing disorders, severe gastrointestinal disorders, major gastrointestinal surgery, or gastric/duodenal ulcers within 6 months prior to screening
* Subject is pregnant, breast feeding, or is of child bearing potential and is not using adequate contraceptive precautions
* Subject is currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug trial(s)
* Subject has experienced a myocardial infarction or major surgery (excluding vascular access surgery) within 3 months prior to screening
* Clinical evidence of current malignancy and/or receiving systemic chemotherapy/radiotherapy with the exception of localized basal cell or squamous cell carcinoma of the skin and cervical intraepithelial neoplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To demonstrate the AMG 223 will produce a statistically significant reduction in serum phosphorus compared with placebo over a 3 week treatment period in subjects with CKD receiving dialysis | TREATMENT PERIOD

SECONDARY OUTCOMES:
To describe a dose response for AMG 223 | TREATMENT PERIOD
To evaluate the safety and tolerability of AMG 223 | ENTIRE STUDY

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com